CLINICAL TRIAL: NCT00646399
Title: A Phase 2b/3, Multi-Center, Randomized, Double-Blind, Placebo Controlled Trial to Evaluate the Safety and Efficacy of Pagibaximab Injection in Very Low Birth Weight (VLBW) Neonates for the Prevention of Staphylococcal Sepsis
Brief Title: Safety and Efficacy of Pagibaximab Injection in Very Low Birth Weight Neonates for Prevention of Staphylococcal Sepsis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biosynexus Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAB-N007
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Results first posted 2011-10-24 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Staphylococcal Sepsis
Keywords: Staphylococcal; Coagulase Negative Staphylococcus; Monoclonal antibodies; Very Low Birth Weight Infants; Prophylaxis
MeSH Terms: interventions — pagibaximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Phosphate Buffered Saline
  Interventions: Drug: Placebo
- Pagibaximab 50 mg/mL (Experimental): Pagibaximab at 100 mg/kg intravenously at Days 0, 1, 2, 9, 16 and 23.
  Interventions: Drug: Pagibaximab 50 mg/mL

INTERVENTIONS:
Drug: Placebo — Phosphate Buffered Saline on Days 0, 1, 2, 9, 16 and 23.
  Arms: Placebo
Drug: Pagibaximab 50 mg/mL — Pagibaximab 100 mg/kg dosed on Days 0, 1, 2, 9, 16 and 23
  Arms: Pagibaximab 50 mg/mL

SUMMARY:
Evaluate the safety, PK and efficacy comparing Pagibaximab Injection to placebo in preventing staphylococcal sepsis in very low birth weight infants. 1550 infants will be enrolled prior to 48 hours of life and will be randomized 1:1 to receive active drug or placebo on study days 0, 1, 2, 9, 16, and 23.

DETAILED DESCRIPTION:
Phase 2b/3, randomized, double-blind, multicenter, placebo-controlled study evaluating the safety, efficacy and pharmacokinetics (PK) of pagibaximab (100 mg/kg/dose) in comparison to placebo for the prevention of staphylococcal sepsis in VLBW infants (600 -1200 grams). Subjects monitored for treatment related adverse events and tolerability to infusion of study drug. Neonatal sepsis will be assessed in the presence of clinical signs and symptoms and one blood culture positive for S. aureus or two blood cultures positive for Coagulase Negative Staphylococci (CoNS). The study period will be 35 days after the first dose or until, death, discharge, or transfer, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. In-patient at a Neonatal Intensive Care Unit (NICU)
2. Informed consent obtained from the legally authorized representative
3. Less than 48 hours old at the time of first infusion
4. Birth weight between 600 grams and 1200 grams
5. Estimated gestation age ≤33 weeks

For multiple gestations, twins may be enrolled if they each meet the entry criteria. They will both be assigned to the same treatment group.

Exclusion Criteria:

1. Infants with history of a hypersensitivity or severe vasomotor reaction to any antibody preparation.
2. Infants with proven staphylococcal infection prior to randomization.
3. Infants with a concomitant infection or other medical condition, whose participation, in the opinion of the Investigator and/or medical advisor, may create an unacceptable additional risk.
4. Immunodeficiency other than due to prematurity.
5. Currently receiving, recently received, or planned to receive other investigational agents that could interfere with conduct or results of this study.
6. Severe congenital or chromosomal anomaly that would limit life expectancy or required corrective measures during the period of this study
7. Uncontrolled seizures

Max Age: 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1579 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Biosynexus Incorporated, Gaithersburg, Maryland, United States

REFERENCES:
- See also: Biosynexus Incorporated — http://www.biosynexus.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 29 Mar 2009 and the last randomized subject completed the trial on 20 Jan 2011. The trial was conducted in the neonatal intensive care unit.
Period: Overall Study
Arm/Group | Pagibaximab | Placebo
Started | 792 | 787
Completed | 709 | 713
Not Completed | 83 | 74
Not completed — Death | 63 | 53
Not completed — Withdrawal by Subject | 9 | 10
Not completed — Other Reason | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pagibaximab | Placebo | Total
Number analyzed (Participants) | 792 | 787 | 1579
Age Continuous [Mean (Standard Deviation); unit: Weeks] — Gestational Age
  Weeks
    600-900g | 25.7 (1.67) | 25.9 (1.83) | 25.8 (1.76)
    901-1200g | 28.0 (1.77) | 27.9 (1.73) | 28.0 (1.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 390 | 393 | 783
  Male | 402 | 394 | 796
Region of Enrollment [Number; unit: participants]
  United States | 603 | 596 | 1199
  Canada | 60 | 59 | 119
  Spain | 54 | 57 | 111
  Italy | 27 | 30 | 57
  United Kingdom | 25 | 28 | 53
  Germany | 23 | 17 | 40
Birth Weight [Number; unit: Participants]
  600-900g | 381 | 371 | 752
  901-1200g | 411 | 416 | 827
Birth Weight [Mean (Standard Deviation); unit: grams]
  600-900g | 758.8 (90.28) | 762.7 (85.05) | 760.7 (87.70)
  901-1200g | 1047.8 (86.25) | 1039.0 (85.72) | 1043.4 (86.05)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Staphylococcal Sepsis From Study Days 0 to 35.
Description: Safety and efficacy
Time Frame: 35 days
Population: 1579 very low birth weight subjects were included in the ITT.
Measure: Number; unit: Participants
Arm/Group | Pagibaximab | Placebo
Number analyzed (Participants) | 792 | 787
Participants | 85 | 79

ADVERSE EVENTS:
Arm/Group | Pagibaximab | Placebo
Serious Adverse Events (participants affected / at risk) | 284/784 | 273/778
Other Adverse Events (participants affected / at risk) | 770/784 | 758/778
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pagibaximab (N=784) | Placebo (N=778)
Necrotizing Colitis (Gastrointestinal disorders) | 52 (52) | 42 (42)
Intraventricular Haemorrhage (Nervous system disorders) | 55 (56) | 57 (58)
Patent Ductus Arteriosus (Congenital, familial and genetic disorders) | 104 (104) | 110 (110)
Intestinal Perforation (Gastrointestinal disorders) | 28 (28) | 26 (28)
Periventricular Leukomalacia (Nervous system disorders) | 14 (14) | 15 (15)
Pulmonary Interstitial Emphysema (Respiratory, thoracic and mediastinal disorders) | 26 (27) | 23 (25)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 12 (12)
Hyperkalaemia (Metabolism and nutrition disorders) | 12 (12) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (18) | 14 (15)
Bradycardia (Cardiac disorders) | 4 (4) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pagibaximab (N=784) | Placebo (N=778)
Anaemia (Blood and lymphatic system disorders) | 479 (646) | 487 (665)
Hypothyroidism (Endocrine disorders) | 9 (9) | 17 (17)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 85 (85) | 79 (79)
Feeding Disorder Neonatal (Metabolism and nutrition disorders) | 204 (221) | 194 (209)
Ophthalmia Neonatorum (Infections and infestations) | 56 (58) | 41 (48)
Cardiac Murmur (Investigations) | 48 (50) | 45 (49)
Hyperbilirubinaemia (Hepatobiliary disorders) | 128 (137) | 112 (113)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other